CLINICAL TRIAL: NCT01017341
Title: PSU Hip Protector for Prevention of Hip Fracture From Falling
Brief Title: Hip Protector for Prevention of Hip Fracture
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Boonsin Tangtrakulwanich, Department of Orthopaedic surgery, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC52-169-11-4-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Hip Fracture
Keywords: hip fracture; back support
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- No hip protector (No Intervention): no hip protector
  Interventions: Device: PSU hip protector

INTERVENTIONS:
Device: PSU hip protector — hip protetor

SUMMARY:
This study aims to evaluate the efficacy of the investigators PSU hip protector for prevention of fracture in elderly.The eligible patients include those with previous diagnosed as unilateral hip fracture. They will be randomized into 2 groups;psu hip protector and no protector. The patients will be instructed to wear the protector fulltime.The inceidence of hip fracture will be compared between both group at the end of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous diagnosed as unilateral hip fracture

Exclusion Criteria:

* Poor communicative ability
* Cannot independently ambulate
* Local skin problem at trocahnteric area

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
incidence of new hip fracture | 6 months, 1 ,2 and 3 yrs

SECONDARY OUTCOMES:
SF 36 | 6 months, 1 ,2 and 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D., Principal Investigator — Department of Othropaedic Surgery, Faculty of Medicine, Prince of Songkla university, Hat Yai, Songkhla,Thailand
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand